CLINICAL TRIAL: NCT06953271
Title: Methenamine Hippurate Compared to Typical Antibiotic Prophylaxis in the Prevention of Urinary Tract Infection Following Intradetrusor OnabotulinumtoxinA Injection for Treatment of Overactive Bladder: a Randomized Controlled Non-Inferiority Trial
Brief Title: Methenamine Hippurate Following Intradetrusor OnabotulinumtoxinA Injection
Acronym: META
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2265134
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Overactive Bladder (OAB); Urinary Tract Infection (Diagnosis)
Keywords: Overactive Bladder; onabotulinumtoxinA; Methenamine; Urinary Tract Infection; BOTOX-A; UTI; OAB
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Tract Infections; Disease | interventions — methenamine hippurate; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Typically prescribed oral antibiotic prophylaxis (Active Comparator): Typically prescribed oral antibiotic prophylaxis for the purposes of this study is defined as oral antibiotics that are routinely prescribed following BOTOX-A injections for UTI prophylaxis. Given known heterogeneity in antibiotic prophylaxis type and duration as well as the lack of standardized antibiotic recommendations for intradetrusor BOTOX-A injections, the choice of antibiotic prophylaxis is deferred to the physician performing the BOTOX-A injections. The duration of treatment will be standardized to three days, based off previous studies.
  Interventions: Drug: Typically prescribed oral antibiotic prophylaxis
- Methenamine hippurate prophylaxis (Experimental): Participants in the experimental arm will receive methenamine hippurate 1 gram by mouth twice daily for three days.
  Interventions: Drug: Methenamine Hippurate

INTERVENTIONS:
Drug: Methenamine Hippurate — Drug: Methenamine hippurate 1 gram by mouth twice daily for three days.
  Arms: Methenamine hippurate prophylaxis
Drug: Typically prescribed oral antibiotic prophylaxis — Drug: typically prescribed oral antibiotic prophylaxis following intradetrusor BOTOX-A injections. This includes, but is not limited to, antibiotic medications such as nitrofurantoin, amoxicillin/clavulanic acid, and trimethoprim/sulfamethoxazole. Dosage will be determined per usual care. Duration of treatment will be standardized to three days.
  Other Names: Oral antibiotics
  Arms: Typically prescribed oral antibiotic prophylaxis

SUMMARY:
The goal of this clinical trial is to compare methenamine hippurate prophylaxis to routine antibiotic prophylaxis following onabotulinumtoxinA (BOTOX-A) injections in women with overactive bladder (OAB). Participants will be randomly selected to receive one of the two post-procedural prophylaxis medications. The primary outcome measure will be urinary tract infection (UTI) rates within 30 days from the BOTOX-A procedure. Secondary outcomes will assess patient satisfaction with the two post-procedural prophylaxis medications.

DETAILED DESCRIPTION:
The purpose of this randomized controlled non-inferiority study is to determine if methenamine hippurate is non-inferior in regards to UTI rate when compared to routinely prescribed antibiotic prophylaxis following intradetrusor BOTOX-A injections for women with OAB. As a secondary aim, this study will also compare patient medication satisfaction, as measured by the Functional Assessment of Chronic Illness Therapy-Treatment Satisfaction-General (FACIT-TS-G) for the two prophylactic medication arms.

Comparators: Methenamine hippurate versus routinely prescribed antibiotic prophylaxis Methenamine hippurate is an oral non-antibiotic antiseptic medication widely used in the prevention of recurrent UTIs.

164 women will be randomly assigned to each treatment option: 82 to methenamine hippurate and 82 to routinely prescribed antibiotic prophylaxis. The primary outcome of UTI rates within 30 days of the BOTOX-A procedure will be calculated for each study arm. The FACIT-TS-G will be administered to participants at the conclusion of the 30-day period.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* undergoing intradetrusor BOTOX-A injections in the office setting for overactive bladder

Exclusion Criteria:

* cisgender male individuals
* neurogenic reasons for bladder symptoms (i.e. spinal cord injury, multiple sclerosis, etc.)
* known allergy and/or contraindication to methenamine hippurate
* currently already taking methenamine hippurate at the time of the procedure
* taking antibiotics for any reason on the day of their BOTOX-A procedure
* positive UTI at time of procedure (positive dip at time of procedure)
* history of bladder cancer
* history of pelvic radiation
* surgically altered detrusor muscle
* pre-procedural need for catheterization
* diagnosis of Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS)
* pregnant or lactating individuals

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Acute Urinary Tract Infection | Date of the BOTOX-A injection to 30 days after the procedure
  Presence of a urinary tract infection (UTI) within 30 days from intradetrusor BOTOX-A injection. UTI will be defined as positive lower urinary tract symptoms (dysuria, hematuria, and/or worsened urinary urgency or frequency) and a positive urine culture.

SECONDARY OUTCOMES:
Medication Satisfaction | Completed over the phone >30 days after BOTOX-A injection.
  We will administer the validated Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction - General (FACIT-TS-G Version 4) survey assessing medication-related (i.e. typical antibiotic or methenamine hippurate) satisfaction and perceived adverse events over the phone >30 days after intradetrusor BOTOX-A injection. The submission of the survey marks the conclusion of the participant's participation in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Sung, MD, MPH, Principal Investigator — Women & Infants Hospital
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tyreman NO, Andersson PO, Kroon L, Orstam S. Urinary tract infection after vaginal surgery. Effect of prophylactic treatment with methenamine hippurate. Acta Obstet Gynecol Scand. 1986;65(7):731-3. doi: 10.3109/00016348609161491. PMID 3544661
- [Background] Schiotz HA, Guttu K. Value of urinary prophylaxis with methenamine in gynecologic surgery. Acta Obstet Gynecol Scand. 2002 Aug;81(8):743-6. doi: 10.1080/j.1600-0412.2002.810810.x. PMID 12174159
- [Background] Davidson SM, Brown JN, Nance CB, Townsend ML. Use of Methenamine for Urinary Tract Infection Prophylaxis: Systematic Review of Recent Evidence. Int Urogynecol J. 2024 Mar;35(3):483-489. doi: 10.1007/s00192-024-05726-2. Epub 2024 Feb 8. PMID 38329493
- [Background] Lee BS, Bhuta T, Simpson JM, Craig JC. Methenamine hippurate for preventing urinary tract infections. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD003265. doi: 10.1002/14651858.CD003265.pub3. PMID 23076896
- [Background] Mouttalib S, Khan S, Castel-Lacanal E, Guillotreau J, De Boissezon X, Malavaud B, Marque P, Rischmann P, Game X. Risk of urinary tract infection after detrusor botulinum toxin A injections for refractory neurogenic detrusor overactivity in patients with no antibiotic treatment. BJU Int. 2010 Dec;106(11):1677-80. doi: 10.1111/j.1464-410X.2010.09435.x. PMID 20590550
- [Background] Shapiro K, Anger J, Cameron AP, Chung D, Daignault-Newton S, Ippolito GM, Lee U, Mourtzinos A, Padmanabhan P, Smith AL, Suskind AM, Tenggardjaja C, Van Til M, Brucker BM. Antibiotic use, best practice statement adherence, and UTI rate for intradetrusor onabotulinumtoxin-A injection for overactive bladder: A multi-institutional collaboration from the SUFU Research Network (SURN). Neurourol Urodyn. 2024 Feb;43(2):407-414. doi: 10.1002/nau.25334. Epub 2023 Nov 30. PMID 38032120
- [Background] Houman J, Moradzadeh A, Patel DN, Asanad K, Anger JT, Eilber KS. What is the ideal antibiotic prophylaxis for intravesically administered Botox injection? A comparison of two different regimens. Int Urogynecol J. 2019 May;30(5):701-704. doi: 10.1007/s00192-018-3721-4. Epub 2018 Aug 3. PMID 30074062
- [Background] Lightner DJ, Wymer K, Sanchez J, Kavoussi L. Best Practice Statement on Urologic Procedures and Antimicrobial Prophylaxis. J Urol. 2020 Feb;203(2):351-356. doi: 10.1097/JU.0000000000000509. Epub 2019 Aug 23. PMID 31441676
- [Background] Getaneh FW, Simhal R, Sholklapper T, Melvin E, Dorris CS, Chou J, Richter LA, Dieter A. Antibiotic prophylaxis for onabotulinum toxin A injections: systematic review and meta-analysis. Int Urogynecol J. 2024 Jan;35(1):19-29. doi: 10.1007/s00192-023-05665-4. Epub 2023 Nov 8. PMID 37938397